CLINICAL TRIAL: NCT05933356
Title: Effectiveness of Exergames on Cognitive, Social Function and Sugar Control Among Chronic Schizophrenia Patients With Diabetes Mellitus in Taiwan
Brief Title: Effectiveness of Exergames on Cognitive, Social Functionamong Chronic Schizophrenia
Acronym: exergames
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KMURCT-SV(I)-20200105
Record Dates: First submitted 2023-05-23; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-05

CONDITIONS: Gambling
Keywords: schizophrenia; cognitive functions; social function; exergames; sugar control
MeSH Terms: conditions — Gambling; Schizophrenia; Social Adjustment

STUDY DESIGN:
Intervention Model Description: Experimental group, in addition to scheduled activities, will be provided with the "individual brain training exergames (a program for improving cognitive function and eye-hand coordination)" three times a week and 30 minutes each time. The control group will be maintained with their scheduled activities in daycare as usual.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group, in addition to scheduled activities, will be provided with the "individual brain training exergames (a program for improving cognitive function and eye-hand coordination)" three times a week and 30 minutes each time.
  "Exergame" and "no intervention" are more informative than "1" and "2"
  Interventions: Behavioral: playing exergames; Other: scheduled activities
- control group (Other): The control group will be maintained with their scheduled activities in daycare as usual.
  Interventions: Other: scheduled activities

INTERVENTIONS:
Behavioral: playing exergames — will be provided with the "individual brain training exergames three times a week and 30 minutes each time
  Arms: Experimental group
Other: scheduled activities — scheduled activities

SUMMARY:
An experimental study with random assignment will be adopted. The participants from 2 hospitals will be assigned to two groups: experimental group (n=77), and control group (n=77). Experimental group, in addition to scheduled activities, will be provided with the "individual brain training exergames (a program for improving cognitive function and eye-hand coordination)" three times a week and 30 minutes each time. The control group will be maintained with their scheduled activities in daycare as usual. Behavioral intentions, cognitive function, social function, and hand-eye coordination will be measured at 0, 3, 6, 9, 12 weeks.

DETAILED DESCRIPTION:
In the first year, an experimental study with random assignment will be adopted. The participants from 2 hospitals will be assigned to two groups: experimental group (n=77), and control group (n=77). Experimental group, in addition to scheduled activities, will be provided with the "individual brain training exergames (a program for improving cognitive function and eye-hand coordination)" three times a week and 30 minutes each time. The control group will be maintained with their scheduled activities in daycare as usual. Behavioral intentions, cognitive function and hand-eye coordination will be measured at 0, 3, 6, 9, 12 weeks.

In the second year, the investigators continue first year study, the experimental group will be provided with the "team cooperation training exergames (a new program for improving sugar control, cognitive and social function)" three times a week and 30 minutes each time. The control group will still be maintained with their scheduled activities in daycare as usual. Cognitive and social function and related physiological indices (muscle mass, fasting blood sugar, glycosylated hemoglobin (HbA1c) and reduction body fat will be measured before intervention and at 0, 3, 6, 9, 12 weeks.

In the third year, in the first three months, the investigators will use the concept of "empowerment" to design a seed program for training 2-3 patients to be "exergame instructors". Experimental group A will be provided with the "team cooperation exergames" three times a week and 30 minutes each time by research team. Experimental group B will be provided with the "team cooperation exergames (teamwork and exercise)" three times a week and 30 minutes each time by "exergame seed ". The control group will be maintained with their scheduled activities in daycare as usual. Cognitive and social function, and related physiological indices will be measured at 0 3, 6, 9, 12 weeks.

The investigators expect this research project can improve the cognitive, social function and sugar control among chronic schizophrenia patients with diabetes mellitus, and the "exergames" can be extended.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia
* aged 20-65 years

Exclusion Criteria:

* Violence or suicidal behavior
* Dementia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Change from MMSEat week 0, 3, 6, 9, and 12.
  Cognitive functions were conducted using the MMSE (Folstein et al., 1975). The MMSE is, in some way, the best known and most widely used measure of cognition in clinical practice worldwide. The MMSE consists of 30 questions for assessing the following seven cognitive domains: orientation in time and place, memory registration and recall, attention and calculation, and language. The total MMSE score ranged from 0 to 30, and higher scores indicate better cognitive functions.
Behavioral intentions | Change from baseline behavioral intentions at week 0, 3, 6, 9, and 12.
  We measured participants' behavioral intention to play exergames using a questionnaire on the behavioral intention, which consisted of four items, and each item used a 5-point Likert scale to assess the levels of agreement with each statement. The contents of this questionnaire were as follows: "In your opinion, will you play and try different exergames in the future? Do you think that exergames can make you relaxed or vigorous?" The total score for the four items ranged from 0 to 16. Higher scores indicate a stronger intention to play exergames. The test-retest (two weeks) intraclass correlation coefficient was 0.88.
One touch' s AC sugar | Change from baseline AC sugar at week 0, 3, 6, 9, and 12.
  One touch' s AC sugar
The Positive and Negative Syndrome Scale (PANSS) | Change from baseline Positive and Negative Syndrome at week 0, 3, 6, 9, and 12.
  The PANSS is among the best-validated instrument for assessing positive, negative, and general psychopathology symptoms associated with schizophrenic patients. It is a standardised clinical interview that rates the presence and severity of positive and negative symptoms, as well as general psychopathology symptoms (e.g., anxiety, depression, etc.) within the past week for schizophrenic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yen Hsueh-Wei, Study Chair — Approval of Clinical Trail/Research
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen HH, Lin CC, Yu ML, Wu HL, Shen HC, Hsieh HF. Active Video Games to Improve Behavioral Intentions and Cognitive Function in Patients With Schizophrenia: Randomized Controlled Trial. JMIR Serious Games. 2025 Oct 1;13:e69116. doi: 10.2196/69116. PMID 41032869